CLINICAL TRIAL: NCT05402475
Title: Online Cognitive Behavioural Therapy (CBT) Intervention for Body Dysmorphic Disorder: Comparison of CBT - Mindfulness to CBT Alone
Brief Title: Online Cognitive Behavioural Therapy Intervention for Body Dysmorphic Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHRF - 02
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Body Dysmorphic Disorder; Body Image Disturbance
Keywords: internet-based intervention with health coaching
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: This is a parallel group randomized clinical trial with two active comparison conditions
Who Masked: Participant
Masking Description: Participant will not be informed about which comparison condition to which she has been assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Online cognitive behavioural therapy with the added components of mindfulness meditation
  Interventions: Behavioral: CBT + Mindfulness
- Active comparator (Active Comparator): Online cognitive behavioural therapy alone
  Interventions: Behavioral: CBT + Mindfulness

INTERVENTIONS:
Behavioral: CBT + Mindfulness — Eight weeks of online CBT intervention combined with mindfulness

SUMMARY:
Body Dysmorphic Disorder (BDD) affects 2.3% of the population and is characterized by excessive concerns with imagined or minor defects in physical appearance. Retrospective outcome studies suggest patients affected by BDD don't typically benefit from surgical treatments while cognitive behaviour therapy (CBT) appears to provide symptom - reducing and distress - reducing benefits. Two different 8-week online CBT approaches to assisting individuals with this disorder are compared: one approach will integrate mindfulness meditation methods (in combination with CBT) and one approach will employ CBT methods without reference to mindfulness meditation.

DETAILED DESCRIPTION:
Body Dysmorphic Disorder (BDD) affects 2.3% of the population and is characterized by excessive concerns with imagined or minor defects in physical appearance. Retrospective outcome studies suggest patients affected by BDD typically do not benefit from surgical treatments while cognitive behaviour therapy (CBT) appears to provide symptom - reducing and distress - reducing benefits. In this study two different 8-week online CBT approaches to assist individuals with this disorder are compared: one approach will integrate mindfulness meditation methods (in combination with CBT) and one approach will employ CBT methods without reference to mindfulness meditation.

The purpose of this comparison is to ascertain whether the inclusions of the two additional intervention modalities, demonstrated effective in other studies, adds to positive outcome effects in this disorder. A primary hypothesis is that the 8 week post-intervention outcomes associated with the CBT-mindfulness approach will show significantly more benefit than the comparison group.

ELIGIBILITY:
Inclusion Criteria: On the Body Dysmorphic Disorder Questionnaire, responses indicating current BDD status; -

Exclusion Criteria: Individuals who are currently receiving weekly structured psychotherapy or who meet DSM-V criteria for severe alcohol/substance use disorder in the past 3 months or demonstrated clinically significant suicidal ideation defined as imminent intent, or attempted suicide in the past 6 months. Individuals of co-morbid diagnoses of borderline personality, schizophrenia, bipolar disorder and/or obsessive compulsive disorder are excluded.

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Body Dysmorphic Disorder Symptom Scale | Baseline, Post-Intervention at 8 weeks following Baseline
  A 55-item scale which asks for presence/absence of symptoms and the degree of severity

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 | Baseline, Post-Intervention at 8 weeks following Baseline
  A 9-item self report scale that asks for symptoms of depression and anxiety

OTHER OUTCOMES:
General Anxiety Disorder - 7 | Baseline, Post-Intervention at 8 weeks following Baseline
  A 7-item self report scale that asks for symptoms of anxiety
Brief Pain Inventory | Baseline, Post-Intervention at 8 weeks following Baseline
  A 11-item self report scale that asks for symptoms of pain experience

CONTACTS AND LOCATIONS:
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Publication of results

REFERENCES:
- [Background] Kuck N, Cafitz L, Burkner PC, Hoppen L, Wilhelm S, Buhlmann U. Body dysmorphic disorder and self-esteem: a meta-analysis. BMC Psychiatry. 2021 Jun 15;21(1):310. doi: 10.1186/s12888-021-03185-3. PMID 34130638
- [Derived] Kerry C, Mann P, Babaei N, Katz J, Pirbaglou M, Ritvo P. Web-Based Therapist-Guided Mindfulness-Based Cognitive Behavioral Therapy for Body Dysmorphic Disorder: Pilot Randomized Controlled Trial. JMIR Ment Health. 2024 Jun 12;11:e55283. doi: 10.2196/55283. PMID 38865704